CLINICAL TRIAL: NCT06675240
Title: Meditative Neurofeedback for Depression
Acronym: MediNF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jyoti Mishra, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MediNF
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Depression Disorders
Keywords: meditation; neurofeedback; rumination; EEG; anxiety; depression
MeSH Terms: conditions — Rumination Syndrome; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MediNF (Experimental): Over 10-sessions participants will engage in a breath-focused meditative practice with frontal brain connectivity neurofeedback provided to enhance performance.
  Interventions: Behavioral: MediNF

INTERVENTIONS:
Behavioral: MediNF — Over 10-sessions participants will engage in a breath-focused meditative practice with frontal brain connectivity neurofeedback provided to enhance performance.

SUMMARY:
The goal of this open-label single-arm study is to test a meditative neurofeedback intervention for depressed mood.

DETAILED DESCRIPTION:
The goal of this open-label single-arm study is to test whether a 10-session meditative neurofeedback intervention significantly alleviates depressive symptons as well as improves secondary outcomes of rumination and mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* moderate depression per PHQ9 symptom ratings

Exclusion Criteria:

* active substance abuse/dependence
* psychotic disorders
* bipolar disorder
* displaying acutely suicidal behaviors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
PHQ9 | 8 weeks
  Depression Symptoms on the Patient Health Questionnaire 9-item (PHQ9) scale, min 0 max 27 with lower scores representing better outcome

SECONDARY OUTCOMES:
MAAS | 8 weeks
  Mindfulness on the Mindful Attention Awareness Scale (MAAS), min 6 max 84 with higher scores representing better outcome
RRQ | 8 weeks
  Rumination on the Ruminative Response Questionnaire (RRQ) scale, min 22 max 88 with lower scores representing better outcome
GAD7 | 8 weeks
  Anxiety symptoms on the Generalized Anxiety Disorder 7-item (GAD7) scale, min 0 max 21 with lower scores representing better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No